CLINICAL TRIAL: NCT01199913
Title: Incidence of Postoperative Cognitive Dysfunction in Elderly Patients Following Desflurane or Sevoflurane General Anesthesia: A Randomized, Controlled Trial
Brief Title: POCD in Elderly Patients Following Desflurane or Sevoflurane General Anesthesia
Status: Completed | Type: Observational
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Richard Applegate, MD, Loma Linda University
Other Study IDs: 5100193
Record Dates: First submitted 2010-09-09; First posted 2010-09-13 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: 1. Postoperative Cognitive Dysfunction
Keywords: problems with thinking after surgery;

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- desflurane and sevoflurane: Subjects will be randomized to either desflurane or sevoflurane. They will be given the Mini Mental State exam at 1, 6 and 24 hours after the end of anesthesia.
  Interventions: Other: The intervention will be Mini-Mental Status Examination (MMSE)

INTERVENTIONS:
Other: The intervention will be Mini-Mental Status Examination (MMSE) — A questionnaire given to the study patient before and after the anesthetic at 1, 6 and 24 hours.

SUMMARY:
The use of desflurane in elderly subjects (>65 years old) undergoing general anesthesia with endotracheal intubation will result in decreased POCD compared to sevoflurane if the patient's MAP is within 20% of the patient's baseline and the cerebral suppression state index stays within the moderately anesthetized range during general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>65 years old)
* Scheduled for elective surgery requiring general anesthesia at LLUMC HSH
* Airway management expected to include endotracheal intubation
* Expected surgical duration 120 to 240 minutes

Exclusion Criteria:

* Pre-existing significant psychiatric disease or mental status changes
* Clinically significant cardiovascular, respiratory, hepatic, renal,neurological, psychiatric, or metabolic disease
* Patient's weighing >50% ideal body weight

  * Men: Ideal Body Weight (in kilograms) = 50 + 2.3 kg per inch over 5 feet
  * Women: Ideal Body Weight (in kilograms) = 45.5 + 2.3kg per inch over 5 feet
* Patients who have undergone a general anesthetic within the past 7 days
* Patient refusal

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Adult patients, male and female, 65 years or older scheduled for elective surgery requiring general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2010-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
POCD in Elderly Patients Following Desflurane or Sevoflurane General Anesthesia | Both groups will complete the MMSE at 1, 6, and 24 hours after the end of anesthesia or to disharge up to 7 days.
  The primary outcome measure will be changes in cognitive function after anesthesia as measured by MMSE.

SECONDARY OUTCOMES:
Secondary outcome measures will include: 1) time to extubation, anesthetic complications (e.g. coughing during extubation), 2) time to readiness for discharge from PACU, 3) length of hospital stay, and 4) any postoperative complications. | 24 hours to 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Loma Linda University, Loma Linda, California, United States

REFERENCES:
- [Derived] Meineke M, Applegate RL 2nd, Rasmussen T, Anderson D, Azer S, Mehdizadeh A, Kim A, Allard M. Cognitive dysfunction following desflurane versus sevoflurane general anesthesia in elderly patients: a randomized controlled trial. Med Gas Res. 2014 Mar 25;4(1):6. doi: 10.1186/2045-9912-4-6. PMID 24666542